CLINICAL TRIAL: NCT03414827
Title: Genetic Evaluation of Renal Cell Carcinoma; Predicting Biomarkers for Renal Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Nessn Azawi, Clinical Professor, Zealand University Hospital
Other Study IDs: SJ-608
Record Dates: First submitted 2018-01-13; First posted 2018-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recruitment of participants to the study takes place at the urological department at Zealand University Hospital, Roskilde, Feb. 2018-April 2018. 10 people with diagnosis of renal cancer should be recruited in phases 1. Subsequently, biological materials from 100 patients with kidney cancer will be used from the national Biobank. In phase 3, 10 patients will be recruited for the final gene test.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with kidney cancer.

Exclusion Criteria:

* Patients without signs of malignancy at final histology report.
* Incapacitated patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients who have been diagnosed with kidney cancer and found suitable for inclusion will be included in the project.
  * The biological material has been collected during routine treatment.
  * Biological material has not been collected in connection with a previous study.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
DNA | 30 days
  Sequence variation in specific genes

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

REFERENCES:
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306